CLINICAL TRIAL: NCT01786330
Title: Do Elastic Abdominal Binders Reduce Post Operative Pain and Blood Loss?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zachary Kuhlmann, DO (Other)
Responsible Party: Sponsor-Investigator, Zachary Kuhlmann, DO, Principal Investigator, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 220121565; 12-049
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Postpartum Hemorrhage; Pain
MeSH Terms: conditions — Postpartum Hemorrhage; Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Group receives elastic abdominal binders after surgery. Binder used is Procare manufactured by DJO, LLC. Binders are to be worn for 24 hours after surgery.
  Interventions: Device: Procare abdominal binder
- Control (Active Comparator): Group receives standard of care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Procare abdominal binder
  Arms: Intervention
Other: Standard of Care
  Arms: Control

SUMMARY:
This is a pilot study investigating the use of abdominal binders after cesarean sections. The researchers are testing whether elastic abdominal binders improve postoperative pain control and reduce postoperative blood loss. Blood loss and pain control are both concerns after giving birth. It is hoped that the use of an abdominal binder after giving birth will provide a non-pharmacologic way to to reduce blood loss and manage pain.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section at term (at least 39 weeks gestation) scheduled in advance
* Singleton gestation confirmed by ultrasound in the current pregnancy
* Body mass index 20-40 kg/m2 (at first prenatal visit or pre-pregnancy)
* None of these pregnancy complications in the current pregnancy:

  1. bleeding disorder or use of anticoagulants other than low-dose heparin
  2. abnormal placenta (placenta previa or accrete)
  3. Preoperative hemoglobin less than 10 mg/dL
  4. Chorioamnionitis (intrauterine infection)
* No chronic pain syndrome (defined as participating in formal chronic pain management within the past year)
* Able to read English and understand spoken English

Exclusion Criteria:

* Onset of labor prior to time when the cesarean was scheduled
* Complications during performance of cesarean or discovered during cesarean:

  1. placenta accreta, increta, or percreta
  2. vasa previa
  3. cesarean hysterectomy required for severe hemorrhage
  4. organ damage during cesarean (cystotomy, enterotomy, ureteral injury)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Kuhlmann, DO, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - Kansas School of Medicine-Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 66 women assessed for eligibility. Of those women, six were excluded from the trial before being assigned to groups. Of the six women excluded: three presented to the hospital in labor prior to the scheduled cesarean, two reported for treatment for chronic pain, and one woman wanted the intervention regardless of randomization.
Groups:
- Intervention: Group receives elastic abdominal binders after surgery. Binder used is Procare manufactured by DJO, LLC. Binders are to be worn for 24 hours after surgery.
  Procare abdominal binder
- Control: Group receives standard of care
  Standard of Care
Period: Overall Study
Arm/Group | Intervention | Control
Started | 30 | 30
Completed | 29 | 27
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Excluded intraoperatively | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (4.7) | 27.7 (4.4) | 28.1 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 27 | 56
Previous vaginal births [Median (Full Range); unit: vaginal births] | 0 [0 to 3] | 0 [0 to 1] | 0 [0 to 3]
Previous cesarean deliveries [Median (Full Range); unit: cesarean deliveries] | 1 [0 to 4] | 1 [0 to 3] | 1 [0 to 4]
Body mass index calculated during 1st visit [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (6.6) | 28.6 (6.3) | 28.7 (6.4)
Gestational age at cesarean delivery [Mean (Standard Deviation); unit: weeks] | 39.1 (0.3) | 39.3 (0.6) | 39.2 (0.5)
Infant birth weight [Mean (Standard Deviation); unit: grams] | 3632.5 (449.2) | 3525.2 (514.8) | 3580.8 (480.6)
Breech presentation [Number; unit: participants] | 3 | 3 | 6
Received epidural [Number; unit: participants] | 28 | 27 | 55
Received Duramorph [Number; unit: participants] | 29 | 27 | 56
Number of pads used during 24 hours postoperative [Mean (Standard Deviation); unit: pads used] | 5.29 (2.27) | 5.48 (1.95) | 5.38 (2.1)

OUTCOME MEASURES:

1. Secondary Outcome: Change in Hemoglobin Concentration
Description: Hemoglobin concentration will be assessed 24 hours after surgery by assessing routine post-operative lab values. Outcome is reported as average difference between pre-operative hemoglobin concentration and post-operative hemoglobin concentration. The negative number indicates the drop in hemoglobin concentration postoperatively.
Time Frame: 24 hours from baseline
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 27
g/dL | -1.84 (1.33) | -1.43 (0.61)

2. Primary Outcome: Lowest Pain Level Postoperative
Description: SF-MPQ2 Pain assessment scale was used to measure lowest pain level postoperative. The pain assessment was self-administered. Lowest pain was reported using a 0 to 10 scale, with 0 being "no pain" and 10 being "pain as bad as you can imagine." Lowest pain level is reported as means for each participant group.
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 27
units on a scale | 1.66 (1.47) | 2.56 (1.22)

3. Primary Outcome: Average Pain Level Postoperative
Description: SF-MPQ2 Pain assessment scale was used to measure average pain level postoperative. The pain assessment was self-administered. Average pain was reported using a 0 to 10 scale, with 0 being "no pain" and 10 being "pain as bad as you can imagine." Reported average pain level is reported as means for each participant group.
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 27
units on a scale | 3.45 (1.74) | 4.48 (1.60)

4. Primary Outcome: Worst Pain Level Postoperative
Description: SF-MPQ2 Pain assessment scale was used to measure worst pain level postoperative. The pain assessment was self-administered. Worst pain was reported using a 0 to 10 scale, with 0 being "no pain" and 10 being "pain as bad as you can imagine." Worst pain level is reported as means for each participant group.
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 29 | 27
units on a scale | 6.41 (2.47) | 6.67 (1.80)

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 2/29 | 0/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=29) | Control (N=27)
Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Extended period of time wearing the abdominal binder resulted in itching.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No